CLINICAL TRIAL: NCT02459834
Title: An Acute Randomized Dose-finding Equivalence Trial of Small, Catalytic Doses of Fructose and Allulose on Postprandial Carbohydrate Metabolism: The Fructose and Allulose Catalytic Effects (FACE) Study
Brief Title: The Fructose and Allulose Catalytic Effects (FACE) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Tate & Lyle (Industry)
Responsible Party: Principal Investigator, John Sievenpiper, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: UT-FACE 2015
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes
Keywords: Allulose; Fructose; Dose Response; Catalytic Dose; Carbohydrate metabolism; Randomized clinical trials
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — psicose; Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Allulose + 75g OGTT (Experimental): Allulose added to a 75 g OGTT of 500 mL at 2 doses (5g and 10g). The drinks will be matched as much as possible in appearance, taste (sweetness), texture, and packaging.
  Interventions: Other: Allulose
- Fructose + 75g OGTT (Experimental): Fructose added to a 75 g OGTT of 500 mL at 2 doses (5g and 10g). The drinks will be matched as much as possible in appearance, taste (sweetness), texture, and packaging.
  Interventions: Other: Fructose
- 75g OGTT (Control) (Active Comparator): A 75 g OGTT (alone) of 500 mL will be given to each participant. The drinks will be matched as much as possible in appearance, taste (sweetness), texture, and packaging.
  Interventions: Other: Control

INTERVENTIONS:
Other: Allulose — A double-blind, randomized, multiple-crossover "equivalence" design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 week washout period. The treatment will be developed by Tate & Lyle.
  Other Names: D-psicose
  Arms: Allulose + 75g OGTT
Other: Fructose — A double-blind, randomized, multiple-crossover "equivalence" design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 week washout period. The treatment will be developed by Tate & Lyle.
  Arms: Fructose + 75g OGTT
Other: Control — A double-blind, randomized, multiple-crossover "equivalence" design. Each participant will act as their own control receiving the treatments in random order, each separated by a 1 week washout period. The treatment will be developed by Tate & Lyle.
  Arms: 75g OGTT (Control)

SUMMARY:
Diabetes remains one of the most important unmet prevention and treatment challenges, and the prevalence of diabetes continues to grow. Some functional food ingredients may hold promise as potential therapies for diabetes. One such functional food is allulose, which is a c-3 epimer of fructose. Allulose is a non-caloric sugar found naturally in small amounts in foods such as dried fruits, brown sugar and maple syrup. Previous research has found that catalytic doses of fructose and allulose have been shown to decrease the postprandial glycemic responses to high glycemic index meals. Fructose, in exchange for other carbohydrates, has also been found to decrease HbA1c levels. Whether the effects of fructose and allulose are equivalent is of particular interest, as allulose represents a non-caloric alternative to fructose. The minimum 'catalytic' dose at which improvements in carbohydrate metabolism are observed also remains to be determined for each of the sugars in people with and without diabetes. This study is an acute randomized controlled dose-finding equivalence trial to assess the effect of fructose and allulose at 2 dose levels (5g and 10g) compared with control (0g) on the glucose and insulin responses to a 75g oral glucose tolerance test (OGTT) in healthy and type 2 diabetes participants.

DETAILED DESCRIPTION:
Diabetes remains one of the most important unmet prevention and treatment challenges. Despite the growing armamentarium of medications, which include six new classes of drugs since metformin was first approved in 1995 in the US, the combined prevalence of impaired glucose tolerance (IGT) and diabetes continues to grow. Although oral antihyperglycaemic agents have been shown to prevent the development of diabetes in high-risk individuals and to reduce the risk of microvascular complications in individuals with type 2 diabetes, they have failed to deliver the anticipated macrovascular benefits.

Some functional food ingredients may hold promise as potential therapies for diabetes. An emerging literature has shown that low-dose fructose and its c-3 epimer, allulose (a non-caloric sugar found naturally in small amounts in foods such as dried fruits, brown sugar, and maple syrup which is generally recognized as safe [GRAS] by the FDA under GRN 400 since 2012 and GRN 498 since 2014) may benefit glycemic control.

Clinical translation of these findings has proven promising. Catalytic doses of fructose at 7.5g and 10g and allulose at 5g, 7.5g, and 10g (but not 2.5g) have been shown to decrease the postprandial glycemic responses to high glycemic index meals (oral glucose, maltodextrins, or mashed potatoes) from ~15-30% in healthy participants and those with prediabetes or diabetes. These acute effects have been shown to be sustainable over the longer term in the case of fructose. In separate systematic reviews and meta-analyses of controlled feeding trials, the investigators showed that both small doses (defined as ≤36g/day based on 3 meals at ≤10g/meal and 2 snacks at ≤3g/snack) and higher doses (median, 60g/day) of fructose in exchange for other carbohydrates decreased HbA1c by 0.4% and 0.53%, respectively, a level of reduction which exceed the clinically meaningful threshold of 0.3% proposed by the Federal Drug Administration (FDA) for the development of new oral anti-hyperglycemic agents.

Although these findings provide a compelling proof of concept, there is an urgent need for replication studies. Whether the effects of fructose and allulose are equivalent is of particular interest, as allulose represents a non-caloric alternative to fructose. The minimum 'catalytic' dose at which improvements in carbohydrate metabolism are observed also remains to be determined for each of the sugars in people with and without diabetes.

OBJECTIVES

* To assess the acute catalytic effects of fructose and allulose at 2 dose levels (5g, 10g) compared with control (0g) on glucose and insulin responses to a 75g oral glucose tolerance test (75g-OGTT) in healthy participants and participants with type 2 diabetes.
* To assess whether there is a dose response or threshold over the proposed dose range (0g, 5g, 10g) for the effects of fructose and allulose on glucose and insulin responses to a 75g-OGTT in healthy participants and participants with type 2 diabetes.
* To assess whether the effects of allulose and fructose are equivalent on the primary endpoint of incremental area under the curve (iAUC) for plasma glucose across the 2 dose levels (5g and 10g) compared with control (0g) in healthy participants and participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants:

  * Adult males and non-pregnant females
  * Normal weight
  * Non-smokers
  * Free of any disease or illness
  * Do not regular take any medications
  * Have a primary care physician
* Diabetes participants:

  * Well-controlled diabetes on diet and/or oral antihyperglycemic agents
  * Not taking insulin
  * Free of any major illness
  * Have a primary care physician

Exclusion Criteria:

* Healthy participants:

  * Age <18 or >75y, Pregnant female
  * Regular medication use
  * Complementary or alternative medicine (CAM) use
  * BMI<18.5kg/m2, >30kg/m2
  * Prediabetes or diabetes (HbA1c≥6%, FBG≥6.1mmol/L)
  * Hypertension (BP≥140/90), Dyslipidemia (Canadian Cardiovascular Society guidelines)
  * Metabolic syndrome (harmonized definition)
  * Polycystic ovarian syndrome
  * Cardiovascular disease
  * Gastrointestinal disease
  * Previous bariatric surgery
  * Liver disease (abnormal liver enzymes)
  * Hyperthyroidism (abnormal TSH)
  * Hypothyroidism (abnormal TSH)
  * Nephropathy (albumin-to-creatinine ratio [ACR] >20)
  * Chronic kidney disease (eGFR >60ml/min/1.73m2)
  * Inflammatory conditions (CRP>3g/L)
  * Acute or chronic infection (abnormal white blood cell count (WBC), CRP>3g/L)
  * Anemia (abnormal Hb)
  * Lung disease
  * Cancer/malignancy
  * Psychiatric illness
  * Major surgery in the last 6 months
  * Other major illness
  * Smoker
  * Heavy alcohol use (>3 drinks/day)
* Diabetes participants:

  * Age <18 or >75y
  * Pregnant female
  * Poorly controlled diabetes (HbA1c>7.5%)
  * Recent diabetes medication change (< 3 months)
  * Insulin use
  * Complementary or alternative medicine (CAM) use
  * BMI<18.5kg/m2, ≥35kg/m2
  * Cardiovascular disease
  * Retinopathy
  * Neuropathy
  * Diabetic foot
  * Gastrointestinal disease
  * Previous bariatric surgery
  * Liver disease (abnormal liver enzymes)
  * Hyperthyroidism (abnormal TSH)
  * Hypothyroidism (abnormal TSH)
  * Anemia (abnormal Hb)
  * Nephropathy (albumin-to-creatinine ratio [ACR] >20)
  * Chronic kidney disease (eGFR >60ml/min/1.73m2)
  * Inflammatory conditions (CRP>3g/L)
  * Acute or chronic infection (abnormal WBC, CRP>3g/L)
  * Lung disease
  * Cancer/malignancy
  * Psychiatric illness
  * Major surgery in the last 6 months
  * Other major illness
  * Smoker
  * Heavy alcohol use (>3 drinks/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Plasma glucose iAUC | up to 12 weeks

SECONDARY OUTCOMES:
Plasma glucose total AUC | up to 12 weeks
Plasma insulin iAUC | up to 12 weeks
Plasma insulin total AUC | up to 12 weeks
Maximum concentrations (Cmax) for plasma glucose and insulin | up to 12 weeks
Time of maximum concentrations (Tmax) for plasma glucose and insulin | up to 12 weeks
Matsuda whole body insulin sensitivity index (Matsuda ISI OGTT); | up to 12 weeks
Early insulin secretion index (∆PI30-0/∆PG30-0); | up to 12 weeks
Insulin secretion-sensitivity index-2 (ISSI-2) | up to 12 weeks
Mean incremental plasma glucose and insulin responses | up to 12 weeks
Mean plasma glucose and insulin responses | up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD PhD FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Sievenpiper JL, de Souza RJ, Cozma AI, Chiavaroli L, Ha V, Mirrahimi A. Fructose vs. glucose and metabolism: do the metabolic differences matter? Curr Opin Lipidol. 2014 Feb;25(1):8-19. doi: 10.1097/MOL.0000000000000042. PMID 24370846
- [Background] Cozma AI, Sievenpiper JL, de Souza RJ, Chiavaroli L, Ha V, Wang DD, Mirrahimi A, Yu ME, Carleton AJ, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Beyene J, Kendall CW, Jenkins DJ. Effect of fructose on glycemic control in diabetes: a systematic review and meta-analysis of controlled feeding trials. Diabetes Care. 2012 Jul;35(7):1611-20. doi: 10.2337/dc12-0073. PMID 22723585
- [Background] Sievenpiper JL, Chiavaroli L, de Souza RJ, Mirrahimi A, Cozma AI, Ha V, Wang DD, Yu ME, Carleton AJ, Beyene J, Di Buono M, Jenkins AL, Leiter LA, Wolever TM, Kendall CW, Jenkins DJ. 'Catalytic' doses of fructose may benefit glycaemic control without harming cardiometabolic risk factors: a small meta-analysis of randomised controlled feeding trials. Br J Nutr. 2012 Aug;108(3):418-23. doi: 10.1017/S000711451200013X. Epub 2012 Feb 21. PMID 22354959
- [Background] Agius L, Peak M. Intracellular binding of glucokinase in hepatocytes and translocation by glucose, fructose and insulin. Biochem J. 1993 Dec 15;296 ( Pt 3)(Pt 3):785-96. doi: 10.1042/bj2960785. PMID 8280078
- [Background] Van Schaftingen E, Detheux M, Veiga da Cunha M. Short-term control of glucokinase activity: role of a regulatory protein. FASEB J. 1994 Apr 1;8(6):414-9. doi: 10.1096/fasebj.8.6.8168691.
- [Background] Hossain MA, Kitagaki S, Nakano D, Nishiyama A, Funamoto Y, Matsunaga T, Tsukamoto I, Yamaguchi F, Kamitori K, Dong Y, Hirata Y, Murao K, Toyoda Y, Tokuda M. Rare sugar D-psicose improves insulin sensitivity and glucose tolerance in type 2 diabetes Otsuka Long-Evans Tokushima Fatty (OLETF) rats. Biochem Biophys Res Commun. 2011 Feb 4;405(1):7-12. doi: 10.1016/j.bbrc.2010.12.091. Epub 2010 Dec 25. PMID 21187061
- [Background] Shiota M, Moore MC, Galassetti P, Monohan M, Neal DW, Shulman GI, Cherrington AD. Inclusion of low amounts of fructose with an intraduodenal glucose load markedly reduces postprandial hyperglycemia and hyperinsulinemia in the conscious dog. Diabetes. 2002 Feb;51(2):469-78. doi: 10.2337/diabetes.51.2.469. PMID 11812757
- [Background] Hawkins M, Gabriely I, Wozniak R, Vilcu C, Shamoon H, Rossetti L. Fructose improves the ability of hyperglycemia per se to regulate glucose production in type 2 diabetes. Diabetes. 2002 Mar;51(3):606-14. doi: 10.2337/diabetes.51.3.606. PMID 11872657
- [Background] Petersen KF, Laurent D, Yu C, Cline GW, Shulman GI. Stimulating effects of low-dose fructose on insulin-stimulated hepatic glycogen synthesis in humans. Diabetes. 2001 Jun;50(6):1263-8. doi: 10.2337/diabetes.50.6.1263. PMID 11375325
- [Background] Moore MC, Cherrington AD, Mann SL, Davis SN. Acute fructose administration decreases the glycemic response to an oral glucose tolerance test in normal adults. J Clin Endocrinol Metab. 2000 Dec;85(12):4515-9. doi: 10.1210/jcem.85.12.7053. PMID 11134101
- [Background] Heacock PM, Hertzler SR, Wolf BW. Fructose prefeeding reduces the glycemic response to a high-glycemic index, starchy food in humans. J Nutr. 2002 Sep;132(9):2601-4. doi: 10.1093/jn/132.9.2601. PMID 12221216
- [Background] Iida T, Kishimoto Y, Yoshikawa Y, Hayashi N, Okuma K, Tohi M, Yagi K, Matsuo T, Izumori K. Acute D-psicose administration decreases the glycemic responses to an oral maltodextrin tolerance test in normal adults. J Nutr Sci Vitaminol (Tokyo). 2008 Dec;54(6):511-4. doi: 10.3177/jnsv.54.511. PMID 19155592
- [Background] Hayashi N, Iida T, Yamada T, Okuma K, Takehara I, Yamamoto T, Yamada K, Tokuda M. Study on the postprandial blood glucose suppression effect of D-psicose in borderline diabetes and the safety of long-term ingestion by normal human subjects. Biosci Biotechnol Biochem. 2010;74(3):510-9. doi: 10.1271/bbb.90707. Epub 2010 Mar 7. PMID 20208358
- [Background] Moore MC, Davis SN, Mann SL, Cherrington AD. Acute fructose administration improves oral glucose tolerance in adults with type 2 diabetes. Diabetes Care. 2001 Nov;24(11):1882-7. doi: 10.2337/diacare.24.11.1882. PMID 11679451
- [Derived] Braunstein CR, Noronha JC, Glenn AJ, Viguiliouk E, Noseworthy R, Khan TA, Au-Yeung F, Blanco Mejia S, Wolever TMS, Josse RG, Kendall CWC, Sievenpiper JL. A Double-Blind, Randomized Controlled, Acute Feeding Equivalence Trial of Small, Catalytic Doses of Fructose and Allulose on Postprandial Blood Glucose Metabolism in Healthy Participants: The Fructose and Allulose Catalytic Effects (FACE) Trial. Nutrients. 2018 Jun 9;10(6):750. doi: 10.3390/nu10060750. PMID 29890724